CLINICAL TRIAL: NCT03960281
Title: Retrospective Assessment of Esthetics and Patient-reported Outcomes of Single Implant Crowns
Brief Title: Assessment of Esthetics and Patient-reported Outcomes of Single Implant Crowns
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Sandra AlTarawneh, Assistant Professor, University of Jordan
Other Study IDs: 2019/182
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Pink and White Esthetic Scores; Patient Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single implant crowns in the anterior maxilla: No drugs to be administered. Patients who have had a single implant crown placed since more than one year in the anterior maxilla (second premolar to second premolar) will be invited for a review session for dental examination and to fill the Oral Health Impact Profile (OHIP) questionnaire.
  Interventions: Other: Regular dental examination

INTERVENTIONS:
Other: Regular dental examination — Regular dental examination, and the patient will be asked to fill a questionnaire

SUMMARY:
The aim of this retrospective study is to perform an assessment of esthetic outcomes of single implants and obtain patient reported outcome measures through the use of a satisfaction questionnaire and the OHIP-14 (Oral Health Impact Profile) questionnaire. Dentists will be performing clinical examination including teeth charting and periodontal charting as well as pink/white esthetic score assessment and these outcomes will be compared to the level of patient satisfaction and patient reported outcomes. The results of this research will add evidence-based data on treatment recommendations for teeth replacement with implants from a patient-centered perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Good oral hygiene
* Single implant crown in the esthetic zone (maxillary 2nd premolar to 2nd premolar)
* Implant crown surrounded by natural teeth
* Implant crown opposed by natural dentition or fixed prostheses
* Implant crown has been installed for at least one year

Exclusion Criteria:

* Presence of active infection around the implant
* Presence of active periodontal disease in the esthetic area.
* Opposing removable prosthesis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had a single implant crown placed more than one year ago in the anterior maxilla (second premolar to second premolar) who fit the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
PES/WES scores of single implant crowns in the anterior maxilla | the single implant crown should be "1 year" to "15 years" in function
  Assessment of pink esthetic score/white esthetic score (PES/WES) scores for implant supported prostheses
OHIP questionnaire patient reported outcome | the single implant crown should be "1 year" to "15 years" in function
  Assessment of patient reported satisfaction with esthetics of implant supported single crowns

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Box VH, Sukotjo C, Knoernschild KL, Campbell SD, Afshari FS. Patient-Reported and Clinical Outcomes of Implant-Supported Fixed Complete Dental Prostheses: A Comparison of Metal-Acrylic, Milled Zirconia, and Retrievable Crown Prostheses. J Oral Implantol. 2018 Feb;44(1):51-61. doi: 10.1563/aaid-joi-D-17-00184. Epub 2017 Nov 1. PMID 29091015
- [Background] Brennan M, Houston F, O'Sullivan M, O'Connell B. Patient satisfaction and oral health-related quality of life outcomes of implant overdentures and fixed complete dentures. Int J Oral Maxillofac Implants. 2010 Jul-Aug;25(4):791-800. PMID 20657876
- [Background] Insua A, Monje A, Wang HL, Inglehart M. Patient-Centered Perspectives and Understanding of Peri-Implantitis. J Periodontol. 2017 Nov;88(11):1153-1162. doi: 10.1902/jop.2017.160796. Epub 2017 May 26. PMID 28548884
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Al Habashneh R, Khader YS, Salameh S. Use of the Arabic version of Oral Health Impact Profile-14 to evaluate the impact of periodontal disease on oral health-related quality of life among Jordanian adults. J Oral Sci. 2012 Mar;54(1):113-20. doi: 10.2334/josnusd.54.113. PMID 22466895